CLINICAL TRIAL: NCT01613807
Title: Phase 4 Humalog® Mix50/50(tm) for the Treatment of Insulin Requiring Gestational Diabetes
Brief Title: Humalog® Mix50/50(tm) as a Treatment for Gestational Diabetes
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sansum Diabetes Research Institute (Other)
Collaborators: Eli Lilly and Company (Industry)
Responsible Party: Principal Investigator, Kristin Castorino, DO, Research Physician, Sansum Diabetes Research Institute
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SDRI 08-01; F3Z-US-X031 (Other: Eli Lilly and Company)
Record Dates: First submitted 2012-06-05; First posted 2012-06-07 (Estimated); Results first posted 2022-06-08 (Actual); Last update posted 2022-06-08 (Actual); Status verified 2022-06

CONDITIONS: Gestational Diabetes Mellitus
Keywords: gestational diabetes mellitus; insulin analogues in pregnancy
MeSH Terms: conditions — Diabetes, Gestational | interventions — Insulin Lispro; Insulin, Long-Acting

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Mix 50/50 (Experimental): Insulin LISPRO: 3 doses of Humalog® Mix50/50™ at mealtime.
  Interventions: Drug: Insulin LISPRO
- Usual insulin regimen (Active Comparator): Usual insulin regimen of insulin, Long-Acting and Insulin: 3 injections of Humalog(r) daily with meals; 3 injections of Humulin N (r) daily on rising, mid-afternoon, and at bedtime
  Interventions: Drug: Insulin, Long-Acting and Insulin

INTERVENTIONS:
Drug: Insulin LISPRO — Humalog® Mix50/50™ [50% insulin lispro protamine suspension and 50% insulin lispro injection, (rDNA origin)], three times daily at mealtime. Dose determined by blood glucose history.
  Other Names: Humalog® Mix50/50™
  Arms: Mix 50/50
Drug: Insulin, Long-Acting and Insulin — Usual insulin regimen: Long-acting insulin three times daily on rising, mid-afternoon, and before bed, and insulin lispro three times daily at mealtime. Doses determined by blood glucose history and carbohydrate content of the meal.
  Other Names: Humalin N(r); Humalog (r)
  Arms: Usual insulin regimen

SUMMARY:
Evaluation of the Safety and Efficacy of Humalog® Mix50/50TM administered as 3 injections daily to Humalog® plus Humulin N® insulin administered as 6 separate injections daily in terms of glucose control for women with Gestational Diabetes.

DETAILED DESCRIPTION:
Controlling hyperglycemia during pregnancy decreases the risk of adverse neonatal and maternal outcomes. Not only must fasting glucose be normalized, but clinical evidence also indicates that controlling postprandial hyperglycemia will significantly reduce the risk of adverse neonatal and maternal outcomes.

Standard therapy to achieve near-normal glycemia in gestational diabetes involves combining intermediate-acting basal (NPH) insulin with rapid-acting insulin (insulin lispro), thereby requiring 6 daily injections. Premixed Humalog® Mix50/50TM has the potential advantage over combination rapid-acting plus NPH insulin because it involves fewer injections, and those injections are associated with mealtime. The potential downside to the premixed formulation is nocturnal hypoglycemia associated with the time lag between the dinner and breakfast dose. This study will evaluate the efficacy and safety of Humalog® Mix50/50TM compared to that of Humalog® plus Humulin N® insulin for the treatment of insulin-requiring patients with gestational diabetes mellitus, while monitoring glucose control, intrauterine growth and assessing pregnancy outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant and at least 13 weeks gestation
* Diagnosed with gestational diabetes mellitus
* Failed diet therapy

Exclusion Criteria:

* <18 years old or over 45 years old
* urine dipstick >2+ protein
* blood pressure >140/80 mmHg
* hematocrit <30%
* refusal to take insulin
* inability to understand instructions or to consent to participate.

Ages: 18 Years to 44 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2008-10; Primary Completion 2010-06 (Actual); Study Completion 2010-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kristin Castorino, DO, Principal Investigator — Sansum Diabetes Research Institute

RESULTS

PARTICIPANT FLOW:
Groups:
- Mix 50/50: Premixed "Mix 50/50" at mealtime, three times per day
  Humalog® Mix50/50™ [50% insulin lispro protamine suspension mixed with 50% insulin lispro injection, (rDNA origin)], given subcutaneously three times daily at mealtime, for a maximum of THREE total insulin injections per day. Dose determined by blood glucose history.
- Control Group: Usual Insulin Regmien: Multiple daily injections:
  3 injections of Humalog(r) daily with meals; AND 3 injections of Humulin N (r) daily on rising, mid-afternoon, and at bedtime
  Long-Acting and Rapid-acting insulin administered as SIX separate injections. Long-acting NPH insulin was given three times daily on rising, mid-afternoon, and before bed, and insulin lispro was administered three times daily at mealtime. Doses determined by blood glucose history and carbohydrate content of the meal.
Period: Overall Study
Arm/Group | Mix 50/50 | Control Group: Usual Insulin Regmien
Started | 20 | 20
Completed | 20 | 20
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Mix 50/50: 3 doses of Mix 50/50 at mealtime
  Insulin LISPRO : Humalog® Mix50/50™ [50% insulin lispro protamine suspension and 50% insulin lispro injection, (rDNA origin)], three times daily at mealtime. Dose determined by blood glucose history.
- Usual Insulin Regimen: 3 injections of Humalog(r) daily with meals; 3 injections of Humulin N (r) daily on rising, mid-afternoon, and at bedtime
  Insulin, Long-Acting and Insulin LISPRO : Long-acting insulin three times daily on rising, mid-afternoon, and before bed, and insulin lispro three times daily at mealtime. Doses determined by blood glucose history and carbohydrate content of the meal.
- Total: Total of all reporting groups
Arm/Group | Mix 50/50 | Usual Insulin Regimen | Total
Number analyzed (Participants) | 20 | 20 | 40
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 1 | 1
  Between 18 and 65 years | 20 | 19 | 39
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 29.6 (4.8) | 33.6 (4.5) | 31.6 (4.65)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 20 | 40
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 20 | 20 | 40

OUTCOME MEASURES:

1. Primary Outcome: Hemoglobin A1C
Description: Compare the efficacy and safety of three daily injections of Humalog® Mix50/50TM to six daily injections of Humalog® and Humulin N® insulin, by hemoglobin A1C.
Time Frame: During Pregnancy (at approximately 28 weeks gestation)
Measure: Mean (Standard Deviation); unit: A1c percent
Arm/Group | Mix 50/50 | Usual Insulin Regimen
Number analyzed (Participants) | 20 | 20
A1c percent | 5.5 (0.3) | 5.6 (0.3)

2. Secondary Outcome: Birthweight of Infant
Description: Birthweight of infant born to mother with gestational diabetes using insulin
Time Frame: End of pregnancy
Measure: Mean (Standard Deviation); unit: grams
Arm/Group | Mix 50/50 | Usual Insulin Regimen
Number analyzed (Participants) | 20 | 20
grams | 3178 (519) | 3375 (419)

ADVERSE EVENTS:
Time Frame: 7 months
Description: During pregnancy and postpartum period
Arm/Group | Mix 50/50 | Usual Insulin Regimen
Serious Adverse Events (participants affected / at risk) | 1/20 | 0/20
Other Adverse Events (participants affected / at risk) | 0/20 | 0/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Mix 50/50 (N=20) | Usual Insulin Regimen (N=20)
Fetal demise, placental abruption (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
Subjects in Humalog 50/50 Mix arm were limited to carbohydrates with meals. They were unable to bolus for carbohydrate-containing snacks.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol (2008-11-24): https://cdn.clinicaltrials.gov/large-docs/07/NCT01613807/Prot_000.pdf